CLINICAL TRIAL: NCT00154609
Title: The Use Tradition Chinese Native Medicine Treats the Osteoporosis Research
Brief Title: Davallia Divaricata BL: The Use of Traditional Chinese Native Medicine for Osteoporosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 930701
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2006-01-23 (Estimated); Status verified 2002-01

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — gu-sui-bu

INTERVENTIONS:
Drug: Gu-Sui-Bu (Davallia Divaricata)

SUMMARY:
We, the investigators at National Taiwan University Hospital, have determined the therapeutic and toxic effects of the traditional herb on the ovariectomized Wistar rat.

The final years will determine its effects on the therapy of women who are over 45 years old and postmenopausal with osteoporosis.

DETAILED DESCRIPTION:
Research of this traditional chinese clinical medicine, Gusuibu, curative effect is planned for three years time. The entire study aims to evaluate the effect of the traditional chinese medicine on postmenopausal osteoporosis as well as the possible side effects on the experimental animal and the human body. All subjects were postmenopausal women with established osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal osteoporosis

Exclusion Criteria:

* Insulin dependent diabetes

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2002-01

PRIMARY OUTCOMES:
The project is aimed to investigate the clinical effects of the water extract of Gu-Sui-Bu from the aspects of animal and clinic studies.

CONTACTS AND LOCATIONS:
Overall Officials: Liu Hwa-Chang, Ph.D, Study Chair — National Taiwan University Medical Center
Locations (1):
- National Taiwan University Medical Center, Taipei, 7, Chung-Shan South Road, Taiwan